CLINICAL TRIAL: NCT02199990
Title: the Study of Propofol or Etomidate Affecting to the Cognitive Function for 1-3 Years Old Children in the 7 Days and 3 Months.
Brief Title: The Effect of Propofol or Etomidate on Cognitive Function for 1-3 Years Old Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guilin Medical University, China (Other)
Responsible Party: Principal Investigator, hong yi Jiang,MD, Professor, chief physician, Guilin Medical University, China
Other Study IDs: 49850254-1
Record Dates: First submitted 2014-07-20; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Anesthesia
Keywords: cognitive function; propofol; etomidate;

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Based on China's guangxi guilin for a hernia operation in 1 to 3 years old preschool children propofol and etomidate on behavioral and cognitive function after intravenous anesthesia in according to beta protein in serum and plasma glutamate (Glutamic acid, Glu) and gamma-aminobutyric acid (Gamma aminobutyric acid, GABA) level of observation, the rapid development period children's cognitive function after anesthesia short-term and long-term change process and its possible mechanism is studied, for the current international debate on "anesthetics effects on developing kids brain nerve" research hot spot in the city of clinical basis and research argument, for pediatric anesthesia clinical safety, provide theoretical basis for the rational use of drugs.

DETAILED DESCRIPTION:
1. by selecting the aged 1 to 3, 100 cases of patients with elective surgery, were randomly divided into the propofol group (P group), the etomidate group (group E), all the 50 cases, healthy age 50 cases of children (blank control group, group C) were studied;
2. the children's intelligence equation of the People's Republic of China neuropsychological test: P, E group of preoperative 1 day before operation, postoperative day 3, 3 months neuropsychological test, observe and evaluate patients POCD is happening; Correspond to the experimental group in the same period in group C, i.e., the first test (1 d) preoperatively, 4 days after the second test (3 d) after operation, 3 months after the third test (3 months), observed and compared with experimental neuropsychological testing of variation;
3. laboratory of brain damage index determination: extract internal jugular venous blood in preoperative and perioperative finish 5 ml, with double antibody immune sandwich enzyme-linked immunosorbent (ELISA) method of determination of serum S - 100 beta protein levels, rapid determination of amino acid analyzer, plasma Glu, GABA levels;
4. statistical analysis: use SPSS13.0 statistical software for children with cognitive function before and after operation and serum S - 100 beta protein and serum Glu, GABA levels change research results should carry on the analysis of variance, P < 0.05 for statistical significance.
5. clear rapid development period of infants receive propofol and etomidate on plasma according to beta protein after intravenous anesthesia and Glu, GABA expression and its relationship between the change of cognitive function and clarify all according to propofol and etomidate intravenous anesthesia on the brain is in rapid development period of infant short-term and long-term postoperative cognitive function and its possible mechanism, the influence of safety for children suffering from anesthesia, and to provide theoretical basis for the rational use of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent; elective laparoscopic hernia repair and appendectomy and other non cardiac operation and Department of cerebral surgery; age 1-3; ASA grade I~II;

Exclusion Criteria:

* Heart, lung, liver, kidney function was abnormal; she has a history of asthma, central nervous system diseases, congenital disorders, hyperactivity, anesthesia operation history; there are factors to evaluate any impact cognitive functions such as language, severe visual and hearing impairment; expected before surgery in patients with delayed extubation; any reason not to cooperate to complete the whole test; perioperative bleeding again; postoperative anesthesia operation; operation time >1h; extubation in patients with delayed; quit by researchers in the process of.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1.Guilin 1-3 years due to hernia surgery to receive propofol or etomidate total intravenous anesthesia in children.
  2.1-3 years old healthy children in 4 kindergartens of different level of teachers in the Guilin city.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The concentration of serum S100 β protein | One hour before anesthesia, one hour after the end of anesthesia.
  Respectively one hour before anesthesia, anesthesia for one hour 5 ml of blood from the jugular vein, serum S100β protein concentration.

SECONDARY OUTCOMES:
Plasma levels of Glutamic acid（Glu) and Gamma-aminobutyric acid（GABA) concentration. | One hour before anesthesia, one hour after the end of anesthesia.
  Respectively one hour before anesthesia, one hour after the end of anesthesia 5 ml of blood from the jugular vein, , plasma Glu, GABA concentration.

OTHER OUTCOMES:
The test results of neuropsychology | One day before the operation, third days after the operation, third months after the operation
  Use of "Chinese children's intelligence equation" for young children tested cognitive function evaluation.The test point in time:One day before the operation, third days after the operation, third months after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Lei xun, MD, Study Director — Guilin Medical University, China
Locations (1):
- Guilin Medical University, Guilin, Guangxi, China